CLINICAL TRIAL: NCT06843473
Title: Prevalence of Weight Related Complications Across Diverse Weight Classifications - A Large Cross-sectional Study in India, Pakistan, Philippines and Vietnam
Brief Title: Prevalence of Weight Related Complications Across Diverse Weight Classifications - A Large Study in India, Pakistan, Philippines and Vietnam
Acronym: WEIGHT DIVERSE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8265; U1111-1308-4250 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Obesity-related Complications
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants will be assessed for obesity-related complications, including measurement of Body Mass Index (BMI)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This study is investigating how common weight related health problems are in people of different weight categories in India, Pakistan, Philippines, and Vietnam. The purpose of the study is to understand the prevalence of weight related health problems in different weight groups. Participants will continue their normal care and will not get any treatment as part of this study; participants will continue receiving any treatments their doctor has prescribed. The study will last for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female aged 18 years or older at the time of signing informed consent.
* Presence of at least one Weight-related complication.

Exclusion Criteria:

* Participants less than 18 years of age at the time of signing informed consent.
* Pregnant women and individuals with recent weight loss due to illness, defined as more than 5 percent (%) weight loss in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be assessed for obesity-related complications, including measurement of Body Mass Index (BMI)
Sampling Method: Non-Probability Sample
Enrollment: 1165 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-10-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Weight-Related Complications Across Different Body Mass Index (BMI) Classes | Upon data collection (Day 1)
  Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (15):
- India (7):
  - Bangalore Diabetes Centre, Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - KGN Diabetes and Endocrinology Centre, Mumbai, Maharashtra
  - AIIMS,Delhi, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences_Delhi, Ansārinagar, New Delhi
  - Endeavour Clinic - Centre of Diabetes and Endocrinology, Bhubaneswar, Odisha
  - IPGME&R and SSKM Hospital, Kolkata, West Bengal
- Pakistan (6):
  - Pakistan Institute of Medical Sciences, Islamabad
  - Aga Khan University Hospital, Karachi
  - National Defence Hospital, Lahore
  - National Hospital Lahore, Lahore
  - Mukhtar A Sheikh Hospital Multan, Multan
  - Peshawar General Hospital, Peshawar
- Asian Hospital and Medical Center, Metro Manila, San Juan, Philippines
- Tam Anh TP. Ho Chi Minh General Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com